CLINICAL TRIAL: NCT03194815
Title: A Randomised Phase II Double-blinded Placebo-controlled Trial of Intravenous Immunoglobulins and Rituximab in Patients with Antibody-associated Psychosis (SINAPPS2)
Brief Title: IVIG and Rituximab in Antibody-associated Psychosis - SINAPPS2
Acronym: SINAPPS2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Alasdair Coles, Revd. Prof. Alasdair Coles, Chief Investigator, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SINAPPS 2
Record Dates: First submitted 2017-02-02; First posted 2017-06-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Psychosis; Autoimmune Encephalitis
Keywords: Psychosis; Immunotherapy; Autoantibodies
MeSH Terms: conditions — Psychotic Disorders; Autoimmune Diseases of the Nervous System | interventions — Immunoglobulins, Intravenous; Saline Solution; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous immunoglobulin and Rituximab (Active Comparator): One cycle of intravenous immunoglobulin (IVIG) 2g/kg over 2-5 days (days 1-5) followed by (b) two infusions of 1g rituximab (the first infusion starting between days 28-35, and the second infusion 14 days later), each with 100mg methylprednisolone.
  Interventions: Drug: Intravenous immunoglobulin; Drug: Rituximab
- Placebo (Placebo Comparator): One cycle of 0.9% saline solution over 2-5 days (days 1-5) followed by (b) two infusions of placebo solution alongside placebo pill - in equal volumes to steroid pre-medication and rituximab.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intravenous immunoglobulin — This is a blood product containing antibodies from thousands of healthy donors.
  Other Names: IVIG; Intratect
  Arms: Intravenous immunoglobulin and Rituximab
Drug: Placebo — This is the control, or sham, treatment
  Other Names: Saline solution
  Arms: Placebo
Drug: Rituximab — Rituximab is a type of biological therapy. It removes B-cells and helps to reduce the inflammation
  Other Names: MabThera
  Arms: Intravenous immunoglobulin and Rituximab

SUMMARY:
A randomised phase II double-blinded placebo-controlled trial designed to explore the utility of immunotherapy for patients with acute psychosis associated with anti-neuronal membranes (NMDA-receptor or Voltage Gated Potassium Channel).

Primary objective: To test the efficacy of immunotherapy (IVIG and rituximab) for patients with acute psychosis associated with anti-neuronal membranes.

Secondary objective: To test safety of immunotherapy (IVIG and rituximab) for patients with acute psychosis associated with anti-neuronal membranes.

DETAILED DESCRIPTION:
Investigators propose a randomised double-blinded placebo-controlled trial to test the hypothesis that immunotherapy is an effective treatment of antibody-associated psychosis, either first episode of psychosis or relapse following previous remission. Immunotherapy for the trial consists of one cycle of intravenous immunoglobulin (IVIG: 2g/kg over days 1-4) followed by two infusions of 1g rituximab (at day 28-35, and then 14 days after the first infusion). The rationale for this regime is that it combines a rapid-action treatment (IVIG) to induce remission with a longer-action therapy (rituximab) to maintain remission. It is based on a protocol where elimination of circulating antibodies is the treatment goal, namely "desensitisation" of potential transplant patients who have multiple anti-HLA antibodies capable of inducing hyperacute rejection and also being tested in various trials on clinicaltrials.gov (NCT00642655, NCT01178216, and NCT01502267). Blinding is required to minimise placebo responses in a trial based on symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Acute psychosis >2 weeks. This may either be first episode or relapse after remission (remission defined as having mild or absent symptoms of psychosis for at least 6 months)
* Serum or CSF neuronal membrane autoantibodies at pathological levels (including NMDAR, LGI1 and other)
* Psychosis symptoms as defined by PANSS ≥4 on at least one of the following items: P1, P2, P3, N1, N4, N6, G5 and G9.

Exclusion Criteria:

* Current episode of psychosis greater than 24 months duration
* Co-existing severe neurological disease
* Evidence of current acute encephalopathy
* Hepatitis or HIV infection, pregnancy
* Contraindications to any trial drug
* Concurrent enrolment in another CTIMP

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to start of symptomatic recovery (symptomatic remission sustained for at least 6 months) | up to 18 months
  remission defined as Positive and Negative Syndrome Scale (PANSS) score 3 or less on PANSS items P1, P2, P3, N1, N4, N6, G5 and G9 sustained for 6 months

SECONDARY OUTCOMES:
Time to first treatment response (whether sustained or not) | up to 18 months
  Treatment response defined as score of 3 or less on each of the following PANSS items: P1, P2, P3, N1, N4, N6, G5, and G9.
Relapse rate | 18 months
  Relapse rate is defined as a score 4 or more on PANSS items P1, P2, P3, N1, N4, N6, G5, and G9.
Number of adverse effects | 18 months
  total number of patient reported adverse effects
Proportion of patients reaching 20% reduction in PANSS total score | 12 months
  20% reduction in the PANSS total score (all PANNS items included)
Proportion of patients reaching 30% reduction in PANSS total score | 12 months
  30% reduction in the PANSS total score (all PANNS items included)
Proportion of patients reaching 40% reduction in PANSS total score | 12 months
  40% reduction in the PANSS total score (all PANNS items included)
Changes in the Clinical Global Impression Scale in Schizophrenia (CGI-Schizophrenia) | 12 months
  Change in CGI-Schizophrenia scores from baseline to month 12
Changes in the Young Mania Rating Scale (YMRS) | 12 months
  Change in YMRS total score from baseline to month 12
Changes in the Antipsychotic Non-Neurological Side-Effects Rating Scale (ANNSERS) | 12 months
  Change in ANNSERS total score from baseline to month 12
Changes in the Brief Assessment of Cognition in Schizophrenia (BACS) | 12 months
  Change in BACS scores from baseline to month 12
Changes in the Global Assessment of Functioning scale (GAF) | 12 months
  Change in the GAF score from baseline to month 12

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair Coles, PhD FRCP, Principal Investigator — University of Cambridge, UK
Locations (10):
- United Kingdom (10):
  - Cambridge University Hospitals NH Foundation Trust, Cambridge
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - NHS Greater Glasgow and Clyde, Glasgow
  - The Walton Centre NHS Foundation Trust, Liverpool
  - University College London Hospitals Nhs Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Salford Royal NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lennox B, Yeeles K, Jones PB, Zandi M, Joyce E, Yu LM, Tomei G, Pollard R, Vincent SA, Shimazaki M, Cairns I, Dowling F, Kabir T, Barnes TRE, Lingford Hughes A, Hosseini AA, Harrower T, Buckley C, Coles A. Intravenous immunoglobulin and rituximab versus placebo treatment of antibody-associated psychosis: study protocol of a randomised phase IIa double-blinded placebo-controlled trial (SINAPPS2). Trials. 2019 Jun 7;20(1):331. doi: 10.1186/s13063-019-3336-1. PMID 31174586
- See also: SINAPPS Group website — http://sinapps.org.uk